CLINICAL TRIAL: NCT02540915
Title: The Pediatric Spine Foundation
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 11-1248
Record Dates: First submitted 2015-08-26; First posted 2015-09-04 (Estimated); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Chest Wall and Spinal Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients 17 years or younger: Standard of Care - Registry. Must have been 11 yrs or under at initial treatment/evaluation.
  Interventions: Other: Standard of Care - Registry

INTERVENTIONS:
Other: Standard of Care - Registry — Standard of Care - Registry

SUMMARY:
The Pediatric Spine Foundation is a registry designed to assist spine surgeons to efficiently identify and track patients with chest wall and spinal disorders.

DETAILED DESCRIPTION:
The Pediatric Spine Foundation is a registry designed to assist spine surgeons to efficiently identify and track patients with chest wall and spinal disorders. The registry allows spine surgeons to participate in retrospective and prospective studies for specific spinal disorders.

ELIGIBILITY:
Inclusion Criteria:

* All patients 17 and under that are being treated at Children's Hospital Colorado Orthopaedic department for a chest wall deformity, spine deformity and/or spinal disorder. However, patients must be/have been 11 or under at their initial treatment/evaluation at Children's Hospital Colorado to be included in this study.

Exclusion Criteria:

* Enrollment in another spine registry

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients 17 and under that are being treated at Children's Hospital Colorado Orthopaedic department for a chest wall deformity, spine deformity and/or spinal disorder.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-11; Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Clinical and radiographic measures for children with chest wall deformity, spine deformity and/or spinal disorder. | Approximately 10 years, recording each clinical and/or surgical visit the patient encounters at Children's Hospital Colorado.
  The registry records data from clinical and surgical visits - evaluation date, demographics, cobb angle, kyphosis, ambulatory status, ECG and ECHO measurements, lab results (HbG, Serum CO2, Albumin, Prealbumin), X-rays, pulmonary function test and O2 saturation, primary diagnosis, comorbidities, prior and current treatment, surgical info (days in ICU, blood loss, type of procedure, position of device, fusion details), and complication details.
  An Early Onset Scoliosis 24-Item Questionnaire is also administered each visit. Questions pertain to general health, pain/discomfort, pulmonary function, transfer, physical function, daily living, energy level, emotion, parental impact, financial impact, and satisfaction. For each category there are 1-3 questions where parents can circle one of the five answer choices that vary in severity grade.
  The primary outcome would be to complete numerous small retrospective cohort studies using the data collected prospectively from the registry.

CONTACTS AND LOCATIONS:
Overall Officials: Sumeet Garg, MD, Principal Investigator — Children's Hopsital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States